CLINICAL TRIAL: NCT03992144
Title: "Prevention of Dry Socket by Means of Single Preoperative Oral Dose of Metronidazole and Amoxicillin Compared to Conventional Therapy"
Brief Title: Prevention of Dry Socket by Means of Single Preoperative Antibiotics Compared to Conventional Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Tahseen Shabbir Khooharo, postgraduate trainee, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Tahseen.S.Khooharo
Record Dates: First submitted 2019-06-13; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Dry Socket
Keywords: dry socket; metronidazole; amoxicillin; lower 3rd molars
MeSH Terms: conditions — Dry Socket | interventions — Amoxicillin; Metronidazole; Benchmarking

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- amoxicillin (Experimental): single preoperative oral 500 mg dose of Amoxicillin before extraction of lower 3rd molar and painkillers after extraction for 1st 48 hours then sos.
  Interventions: Drug: Amoxicillin 500 Mg
- metronidazole (Experimental): single preoperative oral 400 mg dose of metronidazol before extraction of lower 3rd molar and painkillers after extraction for 1st 48 hours then sos.
  Interventions: Drug: metronidazole 400mg
- conventional group (Active Comparator): conventional therapy for prevention of dry socket post operative; 400mg metrinidazol 3 times a day for 5 days 500mg of amooxicillin 2 times a day for 5 days painkiller 48 hours after extraction then sos
  Interventions: Drug: metronidazol 400mg and amoxicillin 500mg

INTERVENTIONS:
Drug: Amoxicillin 500 Mg — Amoxicillin 500mg an hour before tooth extraction
  Other Names: amoxill 500mg
  Arms: amoxicillin
Drug: metronidazole 400mg — 400mg of metronidazole an hour before extraction
  Other Names: flygel 400mg
  Arms: metronidazole
Drug: metronidazol 400mg and amoxicillin 500mg — 400mg metronidazole TDS, amoxicillin 500mg BD for 5 days after extraction
  Arms: conventional group

SUMMARY:
Background: One of the commonest post-operative complications after tooth extraction is dry socket; it can be defined as postoperative pain in and around the tooth extraction site, which increases in severity at any time between 3rd to 5th post-operative days along with disintegrated blood clot within the tooth extraction socket with or without halitosis. The exact etiology is unclear therefor prevention remains the main beneficial therapy. Various factors are thought to play an important role in etiology of dry socket including, anaerobes, fibrinolysis, traumatic extractions, frequent spiting and rinsing, oral contraceptive pill and smoking.

Numerous approaches have been tried for prevention of dry socket; include antiseptic mouthwashes, anti-fibrinolytic agents, antibiotics, intra-socket dressings and medicated packing into the extraction wound for example chlorohexidine mouthwashes, warm saline rinses, gelatin sponges, occlusive dressings and oxidized cellulose sponge.

Purpose of the study is to compare the role of single preoperative oral dose of metronidazole with amoxicillin in hindrance of dry socket compared to conventional therapy after removal of mandibular third molar of class 2 impaction.

Objectives: To find out effective treatment for prevention of dry socket among preoperative single oral dose of metronidazole and amoxicillin compared to conventional therapy.

Methods: A double blind randomized control trial in which patients requiring surgical extraction of lower 3rd molar of class 2 impactions were selected for this study. Patients were randomly divided into 3 groups, one of the groups had received single preoperative oral dose of metronidazole one hour before extraction, second group was treated with single oral dose of amoxicillin an hour before tooth extraction and third group was treated with conventional therapy. Patients were asked to visit on 5th postoperative day or before it in case the pain persist or reoccur.

DETAILED DESCRIPTION:
Background Dry socket is one of the commonest problems that occur after extraction of molars. It can be described as a painful inflammatory condition that occurs due to non-formation or early displacement of a blood clot from a tooth extraction site before the healing of wound occurs. Clinical presentation of dry socket is intense ache, bad breath, hollow socket due to displacement of blood clot and exposure of bone. Pain produced by dry socket is known to last from 7 to 14 days. Incidence of dry socket is approximately 3% for routine extractions and can go beyond 30% for impacted lower third molars.

Tooth impaction is a pathological condition in which a tooth fails to erupt to the occlusal level of its normal position. Lower third molars are the most commonly impacted teeth. The prevalence of third molar impaction ranges from 16.7% to 68.6%.

Multiple factors are associated with dry socket formation. such as patient's age, Gender, extraction in posterior region of mouth, smoking status, oral contraceptive.

Incidence of dry socket perhaps lies somewhere from 5% to 20% worldwide.It ranges broadly between 0.9% and 21% in United Kingdom and 3.5% in Siri-Lankan. Incidence of dry socket in Pakistani population is reported 13.8%20.

Incidence of dry socket after extraction of impacted third molars is about 25-30%33.

Third molar is the most frequently impacted tooth and its prevalence ranges from 16.7% to 68.6%.

Methods Data collection was done from the patients requiring surgical extraction of mandibular third molars class two impaction, at outpatient department of oral and maxillofacial department of Dow university health sciences.

Patients were selected according to the inclusion and exclusion criteria. After explaining the purpose of the study and its associated benefits and risks, consent was obtained from the patients. Patients were randomly divided into 3 groups. Ethical approval was obtained from institutional review board of DUHS, Karachi.

Lower 3rd molars with class 2 impaction, both genders, aged between 18 to 40 years were included in the trail. Whereas smokers, alcoholic patients, pregnant and nursing mothers, those taking anticoagulant, oral contraceptives, already taking antibiotics, with renal or hepatic dysfunction, allergic to antibiotics and reluctant to participate were excluded from the trail.

All of the patients were operated by R2 postgraduate trainee of oral and maxillofacial surgery department, under local anesthesia, inferior alveolar and long buccal nerves were anesthetized. Incision was given, flap was elevated and osteotomy and/or tooth section was done depending on the case. Round and fissured burs were used to remove the bone with low speed micrometer straight hand piece. Normal saline was used as coolant and irrigating solution. After extraction of the tooth, socket was irrigated and flushed with normal saline. Sutures were given with 3-0 silk material and a roll of sanitized gauze was placed over the extraction socket and patients were asked to bite on it for at least 40 minutes. prescribed. Post-operative instructions were given to the patients both verbally as well as in written form. On fifth post-operative day patients were examined with naked eye under the light of dental unite. Those diagnosed with dry socket were treated with alveogel after irrigating and flushing the socket with normal saline.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring surgical extraction of lower third molars with class 2 impaction.
* Males and females were included.
* Age range of the patients was between 18 to 40 years.
* Exclusion Criteria:
* Non-surgical extractions, extractions of other then lower molars,
* Infected tooth.
* tooth with grade 3 or greater mobility.
* Reluctant to participate.
* Pregnant ladies.
* Nursing mothers.
* Alcoholic patients.
* Smokers.
* Patients taking oral contraceptives.
* Patient already taking antibiotics.
* Allergic to amoxicillin and metronidazole.
* Patients on anticoagulant therapy i.e. warfarin, nicoumalone, phenytoin, fluocil.
* Those with severe renal and hepatic dysfunction.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
dry socket | 5 days
  Characteristic of interest: patient complaining of moderate to severe pain in or around the tooth extraction site between 3 to 5 post-operative days.
  Measuring instruments: The observation will be performed with naked eye under the light of dental unit and cheek will be retracted via dental mirror instrument.
  Method of testing: Presence of moderate to severe pain, total or incomplete loss of blood clot, bare bone in the socket, and halitosis.
  Decision criteria: Presence of above features at the site of tooth extraction will indicate the presence of dry socket.

CONTACTS AND LOCATIONS:
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan